CLINICAL TRIAL: NCT01732952
Title: Dyslipidemia International Survey - China
Brief Title: Dyslipidemia International Survey-China
Acronym: DYSIS-China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Society of Cardiology (Other)
Responsible Party: Principal Investigator, Hu Dayi, Chinese Society of Cardiology, Chinese Society of Cardiology
Other Study IDs: 0000-271-0
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-11

CONDITIONS: the Prevalence,Lipid Abnormalities,
Keywords: the prevalence,lipid abnormalities,CV risks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- regions,hospitals,age, gender, risk levels, comorbidity,

SUMMARY:
This cross-sectional, non-interventional, and observational study will assess the lipid profile of patients who have been taking lipid-modifying drugs (i.e., proportion of patients achieving treatment to goal according to national and international lipid management guidelines) during a single visit to their physicians on an outpatient basis in 6 representative geo-economic regions in China: Northeast, North, East, South, Southwest, and Northwest; and within each region, in three tiers of hospitals: tier 3 (primary or teaching hospitals), tier 2 (secondary or city level hospitals), and tier 1 (community hospitals/health centers). The investigators will primarily be cardiologists, endocrinologists, neurologists, gerontologists, internists, or other physicians who are representative of the general population of physicians managing patients with dyslipidemia and/or at high risk for cardiovascular events likely to be treated with lipid-modifying drugs. Demographic data, cardiovascular risk factors, a history of cardiovascular disease and cardiovascular treatments will be documented in a single visit through patient clinical examination and chart review.

DYSIS-China is part of a string of epidemiological studies that share the same master protocol, which has been conducted in different countries mainly in Europe and Canada. The analysis of the pooled studies including overall data and cross-country comparisons is the subject of a distinct protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an outpatient > 45 years of age
2. Patient is currently* treated with a statin
3. Patient has a documented fasting lipid profile (> 1 lipid parameter within the last 12 months) performed while on lipid-modifying therapy for at least 3 months
4. Patient agrees to participate in the study by giving informed consent.

   * Patient is already being treated with a lipid-modifying drug just before the visit. Patient for whom a lipid-modifying therapy is initiated at the time of the visit must not be included.

Exclusion Criteria:

1. Patient is currently participating in a clinical trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patient is an outpatient > 45 years of age
  2. Patient is currently* treated with a statin
  3. Patient has a documented fasting lipid profile (> 1 lipid parameter within the last 12 months) performed while on lipid-modifying therapy for at least 3 months
  4. Patient agrees to participate in the study by giving informed consent.
     * Patient is already being treated with a lipid-modifying drug just before the visit. Patient for whom a lipid-modifying therapy is initiated at the time of the visit must not be included.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the prevalence and types of persistent lipid abnormalities in patients aged > 45 years treated with a lipid-modifying drug | 6 months

SECONDARY OUTCOMES:
assess patient characteristics, including CV risk levels, in the subsets of patients with persistent lipid abnormalities | 6months

OTHER OUTCOMES:
explore a potential relationship between the persistence of lipid abnormalities and the local known (historical) prevalence of CV morbidity/mortality | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Hu da yi, Dr., Principal Investigator — Chinese Society of Cardiology
Locations (1):
- Peiking University People' Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen Y, Yin C, Li Q, Yu L, Zhu L, Hu D, Sun Y. Misuse of Aspirin and Associated Factors for the Primary Prevention of Cardiovascular Disease. Front Cardiovasc Med. 2021 Sep 3;8:720113. doi: 10.3389/fcvm.2021.720113. eCollection 2021. PMID 34540919
- [Derived] Yan X, Li Y, Dong Y, Wu Y, Li J, Bian R, Hu D. Blood pressure and low-density lipoprotein cholesterol control status in Chinese hypertensive dyslipidemia patients during lipid-lowering therapy. Lipids Health Dis. 2019 Jan 29;18(1):32. doi: 10.1186/s12944-019-0974-y. PMID 30696435